CLINICAL TRIAL: NCT01064492
Title: A Phase 1, Cross-Over, Single-Dose, Open-Label Study To Estimate The Relative Bioavailability And Food Effect Of PF-04620110 In Healthy Adult Subjects
Brief Title: A Phase 1 Study To Estimate The Relative Bioavailability And Food Effect Of PF-04620110 In Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B0961004
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — PF-04620110

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABC, ACB, BAC, BCA, CAB, and CBA (Experimental)
  Interventions: Drug: PF-04620110

INTERVENTIONS:
Drug: PF-04620110 — The three treatments are A) a single dose of 5 mg PIC under fasted condition; B) a single dose of 5 mg tablet under fasted condition: and C) a single dose of 5 mg tablet under fed condition.

SUMMARY:
PF 04620110 is an acylCoA:diacylglycerol acyltransferase 1 (DGAT1) inhibitor that is being developed for the treatment of type 2 diabetes mellitus (T2DM). It is anticipated that PF 04620110 will have anti diabetic effects through inhibition of intestinal triglyceride absorption and potentially weight loss. The primary purpose of this study is to evaluate the pharmacokinetics, safety and tolerability of multiple oral formulations of PF 04620110 administered to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 lead ECG and clinical laboratory tests).
* Women must be of non childbearing potential.
* Body Mass Index (BMI) of 17.5 to 35.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Endpoints: Cmax, Tmax, AUClast, AUCinf, and half life, as the data permit. | following each treatment

SECONDARY OUTCOMES:
Safety Endpoints: Safety and tolerability of PF 04620110 will be assessed by physical examinations, adverse event monitoring, 12 lead ECGs, vital sign, and clinical safety laboratory measurements. | before, during, and following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0961004&StudyName=A%20Phase%201%20Study%20To%20Estimate%20The%20Relative%20Bioavailability%20And%20Food%20Effect%20Of%20PF-04620110%20In%20Healthy%20Adult%20Subjects%20